CLINICAL TRIAL: NCT06190158
Title: Subclinical Primary Aldosteronism in Diabetes At-Risk for Kidney Disease
Acronym: SubPA-DKD
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Anand Vaidya, Associate Professor, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023p003466
Record Dates: First submitted 2023-12-18; First posted 2024-01-05 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes; Chronic Kidney Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: This is a mechanistic study involving dietary and hormonal interventions to evaluate hormone physiology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- type 2 diabetes at risk for chronic kidney disease (Experimental): type 2 diabetes at risk for chronic kidney disease
  Interventions: Diagnostic Test: Oral sodium suppression test; Diagnostic Test: Saline suppression test; Diagnostic Test: Captopril suppression test; Diagnostic Test: Dexamethasone suppression test; Diagnostic Test: Cosyntropin stimulation test

INTERVENTIONS:
Diagnostic Test: Oral sodium suppression test — Oral sodium suppression test (~2 grams of supplemental sodium for 3 days)
Diagnostic Test: Saline suppression test — Saline suppression test (2 liters of saline)
Diagnostic Test: Captopril suppression test — Captopril suppression test (50mg of captopril)
Diagnostic Test: Dexamethasone suppression test — 1mg of dexamethasone
Diagnostic Test: Cosyntropin stimulation test — 250mcg of cosyntropin

SUMMARY:
The aim of this protocol is to assess the presence and severity of primary aldosteronism pathophysiology in patients with type 2 diabetes who have, or are at-risk for developing, chronic kidney disease.

DETAILED DESCRIPTION:
Diabetes is the leading cause of chronic kidney disease (CKD). When combined, diabetes with CKD exponentially increases risk for cardiovascular disease (CVD) and death. Preventing or delaying CKD in diabetes would substantially decrease these adverse outcomes, save billions in healthcare expenditures, and improve quality of life for those at high-risk for dialysis-dependent kidney failure.

Emerging evidence strongly suggests that primary aldosteronism (PA) pathophysiology is a causative mechanism for the development and progression of CKD in diabetes. PA pathophysiology is characterized by relatively non-suppressible and renin-independent aldosterone production that causes excessive activation of the mineralocorticoid receptor (MR). This maladaptive activation of the MR induces inflammation and fibrosis that contributes to hypertension (HTN), CKD, cardiovascular disease, and death.

PA has traditionally been considered to be a rare and categorical disorder. However, it has been shown that PA pathophysiology exists across a broad continuum of severity, from mild (or subclinical) to overt (or severe); in this regard, PA is better considered to be a pathophysiologic syndrome. The origins of PA pathophysiology can be observed in normotensive and pre-hypertensive people, which consequently increases the risk for developing HTN, developing CKD and progression of CKD to end-stage kidney disease, structural heart disease, and adverse CVD outcomes. Thus, early identification of PA pathophysiology is of critical importance since widely available targeted therapies (such as MR antagonists) can mitigate these adverse outcomes.

The prevalence of PA pathophysiology is high and almost entirely unrecognized. It can be detected in 10-25% of the general population. In high-risk populations, such as those with resistant hypertension and/or hypertension with hypokalemia, the prevalence of PA exceeds 25%. However, despite this alarming prevalence, the rates of testing for PA, or empiric MR antagonist use, in these high-risk populations is abysmal and rarely exceeds 2%. The scope of this problem is magnified by the fact that randomized clinical trials have established the exceptional efficacy of MR antagonists. Landmark trials have established the efficacy of MR antagonist therapy for treating PA, controlling resistant HTN, reducing adverse outcomes in heart failure, reducing albuminuria, and most germane to this proposal, for lowering the risk of CKD progression and incident end-stage kidney disease in patients with diabetes and incident CVD outcomes despite the use of ACEi/ARBs.

GAPS IN CURRENT UNDERSTANDING: What is the mechanism by which MR antagonists impart reno-protective benefits in patients with type 2 diabetes? Ground-breaking results of clinical trials led to the FDA approval of the MR antagonist finerenone and changes to clinical practice guidelines to employ MR antagonists to prevent CKD progression in type 2 diabetes; however, the role of PA pathophysiology was not directly investigated. The investigators hypothesize that there is a prevalent, progressive, and unrecognized, spectrum of PA pathophysiology and MR activation in people with diabetes who have, or are vulnerable to developing, CKD.

The aim of this protocol is to assess the presence and severity of primary aldosteronism pathophysiology in patients with type 2 diabetes who have, or are at-risk for developing, chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years
2. Known diagnosis of type 2 diabetes; or unknown/unclear diagnosis of type 2 diabetes but hemoglobin A1c 5.7-6.4% on screening while on treatment with metformin or SGLT2 inhibitor or GLP1RA class of medications; or unknown/unclear diagnosis of type 2 diabetes but hemoglobin A1c 6.5-8.9% on screening.
3. One of the two following inclusion criteria i. At-risk for developing CKD: eGFR 60-89 mL/min/1.73m2 plus at least one of the following:

   * Moderate albuminuria (30-300 mg/g)
   * Diagnosis of hypertension or active treatment with anti-hypertensive medications
   * BMI ≥ 30 kg/m2 ii. At-risk for CKD progression: eGFR 45-60 mL/min/1.73m2

Exclusion Criteria:

* Type 1 or Type 3 diabetes
* Hemoglobin A1c ≥ 9%
* Inability to safely participate in fasting study visits (determination at the discretion of PI and MD study staff based on cumulative assessment of safety factors)
* Average blood pressure at screening visit of >150 mmHg systolic or >100 mmHg diastolic
* Screening average systolic blood pressure less than 105 mmHg without the use of an ACE inhibitor or angiotensin receptor blocker
* Inability to safely withdraw ACE inhibitor or angiotensin receptor blocker medication in lieu of alternative medication for a few weeks (determination at the discretion of PI and MD study staff based on cumulative assessment of factors)
* Known history of stroke, symptomatic coronary artery disease, myocardial infarction, heart failure, cerebral or aortic aneurysm.
* Known cardiac murmur suggestive of aortic stenosis or mitral regurgitation, or detected newly on screening physical examination
* Active cancer that is being treated with chemotherapeutic agents
* Pregnancy
* Breast feeding
* Daily use of prescribed opioid medications
* Illicit drug use (cocaine, heroin, methamphetamine)
* Daily use of oral glucocorticoids
* Electrocardiogram that shows evidence of prior myocardial infarction, atrial arrhythmia, left or right bundle branch blocks.
* Hematocrit < 32% or Hemoglobin < 10 g/dl (women) or Hemoglobin < 11 g/dl (men) on the day of screening
* eGFR <45 mL/min/1.73m2 on the day of screening
* Known allergy to ACE inhibitors, cosyntropin
* Active use of a mineralocorticoid receptor antagonist

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
The magnitude of non-suppressible and renin-independent aldosterone production following saline suppression | 5 years
  The plasma aldosterone concentration following saline suppression testing will serve as a metric quantifying the degree of renin-independent aldosterone production (PA pathophysiology)
The magnitude of non-suppressible and renin-independent aldosterone production following oral sodium suppression. | 5 years
  The magnitude of non-suppressible and renin-independent aldosterone production measured by urinary aldosterone following oral sodium loading,

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided